CLINICAL TRIAL: NCT00575835
Title: Oral Vitamin D Supplementation in Elderly Women: Twice a Day or Three Times a Year? A Randomised Controlled Trial
Brief Title: Oral Vitamin D Supplementation in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Päivikki and Sakari Sohlberg Foundation, Finland (Other); Lilly Foundation (Unknown)
Responsible Party: Matti Välimäki, MD, Ph.D, Helsinki University Central Hospital, Department of Medicine, Division of Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77/2006
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Optimal Vitamin D Administration
Keywords: vitamin D; seasonal variation; PTH; bone markers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: vitamin D twice daily
- 2 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 oil three times in a year

INTERVENTIONS:
Dietary Supplement: vitamin D twice daily — Kalsipos-D, vitamin D3 400 ID/tbl, 2 tbl/day for one year
  Arms: 1
Dietary Supplement: Vitamin D3 oil three times in a year — Vigantol oil , D3 20000IU/ml, 4.9 ml every four months for one year
  Arms: 2

SUMMARY:
The aim of this study is to compare oral vitamin D supplementation administered in two different ways, namely either twice a day (800IU/d, 292000IU/y) or three times a year (97333IU every 4 months, 292000IU/y) in elderly women in combination with daily supplementation of calcium 1 gram. We will 1)compare the blood concentrations of 25 OH vitamin D in the two treatment groups amd monitor if a sufficient and safe concentration of 25OH D in blood can be maintained with these two treatments.2) Find out seasonal variation in vitamin D concentrations in these treatments. 3) Find out safety of these treatments

ELIGIBILITY:
Inclusion Criteria:

* Females
* 70-80 years
* Living in the community

Exclusion Criteria:

* Renal disease
* Diseases that contraindicate vitamin D supplementation
* Medications affecting bone
* Malignancy

Ages: 70 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Blood 25 OH D vitamin concentrations | 8 times during the year

SECONDARY OUTCOMES:
serum calcium, 24-hour calcium excretion in urine, creatinine clearance | 8 times during the year

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, department of medicine, division of endocrinology, Helsinki, Finland